CLINICAL TRIAL: NCT02879903
Title: Prevalence of Porphyromonas Gingivalis Fimbrial Subunit Genotype in Smokers and Nonsmokers After Periodontal Therapy
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Universidade Federal Fluminense (Other)
Responsible Party: Principal Investigator, Gabriela Alessandra da Cruz Galhardo Camargo, Professor, Universidade Federal Fluminense
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Diagnostic
Other Study IDs: CAAE: 53022216.0.0000.5626
Record Dates: First submitted 2016-08-10; First posted 2016-08-26 (Estimated); Last update posted 2016-08-30 (Estimated); Status verified 2016-08

CONDITIONS: Chronic Periodontitis
Keywords: Porphyromonas gingivalis; Periodontal treatment; Smokers
MeSH Terms: conditions — Chronic Periodontitis | interventions — Periodontal Index; Surveys and Questionnaires

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- biofilm tobacco effect (Experimental): Group smokers - patients will receive periodontal treatment and biofilm will be collected.
  Interventions: Procedure: Periodontal treatment; Procedure: Microbiological collect; Procedure: Questionnaire
- biofilm non smoker effect (Experimental): Group Non Smokers - patients will receive periodontal treatment and biofilm will be collected.
  Interventions: Procedure: Periodontal treatment; Procedure: Microbiological collect; Procedure: Questionnaire

INTERVENTIONS:
Procedure: Periodontal treatment — An experienced periodontist will be performed clinical periodontal parameters, including Plaque Index, Bleeding On Probe, Pocket Probing Depth, Gingival Recession, Clinical Attachment Level using a periodontal probe, at six sites per tooth at all teeth, excluding third molars.
  Quadrant scaling and root planning will be weekly performed on each patient under local anesthesia using periodontal curettes and ultrasonic scalers. The maintenance therapy will be included professional plaque control and Scaling and root planing in recurrent periodontal pockets.
Procedure: Microbiological collect — Biofilm will be collected with the paper point to analyse presence of Porphyromonas gingivalis fimbrial subunit gene type I, II, III, IV and V.
Procedure: Questionnaire — Age will be expressed in years Sex -female and male, will be expressed in percentage. Time of cigarette consumption - will be expressed in years

SUMMARY:
The aims of the present study will be identify 5 types of fimbrial subunit genotype strains in smokers and nonsmokers with periodontitis, before and after periodontal therapy. Third two periodontitis patients will be selected to these study, 16 nonsmokers and 16 smokers. Clinical and microbiological parameters were evaluated at baseline and 3 months after periodontal treatment: Plaque Index, Bleeding On Probe, Probing Depth, Gingival Recession and Clinical Attachment Level. The prevalence of P. gingivalis and fimbrial subunit gene strains will be determined by Polymerase Chain Reaction.

DETAILED DESCRIPTION:
Porphyromonas gingivalis is one of the most prevalent periodontopathogens present in red complex that is considered to be infectious agent causing several types of periodontal diseases. P. gingivalis has ability to invade gingival epithelial cells and can survive for extended periods of time. Fimbriae have been characterized to be key factors in adhesion, invasion, and colonization. Fimbriae are also responsible for invasion of membrane vesicles into host cells. Long fimbriae (FimA), also known as major fimbriae, are long, peritrichous, filamentous components. They have a role in initial attachment and organization of biofilms, as they act as adhesins that mediate invasion and colonization of host cells contributing to P. gingivalis virulence.

Fimbrillin (FimA; structural subunit protein of fimbriae) is classified into 5 variants (types I to V) based on their nucleotide sequences. P. gingivalis strains possessing type II fimA are correlated with P. gingivalis-positive patients, and its occurrence was significantly increased with the more severe forms of periodontitis. Previous studies evaluated the differences among the prevalence of fimA genotypes and periodontal health status in adults. P. gingivalis was detected in 36.8% of the healthy subjects and in 87.1% periodontitis patients. Among the P. gingivalis-positive healthy adults, the most prevalent fimA type was type I (76.1%), followed by type V (29.7%). In contrast, a majority of the periodontitis patients carried type II fimA organisms (66.1%), followed by type IV (28.9%). These findings indicate that there are both disease-associated and non-disease-associated strains of P. gingivalis, and that their infectious traits influencing periodontal health status could be differentiated based on the clonal variation of fimA genes.

Tobacco consumption is a risk factor for periodontal disease. Several studies have been reported that smoker habit is associated with greater clinical attachment loss, recession and tooth loss and reduced bone height and density. However, controversial report has been discussed about the differences between smokers and non-smokers periodontopathogens. P. gingivalis have been report 52.2% prevalence in non-smokers and 66.7% in smokers (pocket depth 3-5 mm) , and are associated with high levels in sites with periodontitis.

The mechanism that tobacco affects the periodontal tissue is related with nicotine that has been associated with various cellular changes that may contribute to the initiation and subsequent progression of periodontal disease. It is promote local effect like the reduction of the gingival blood flow, what can be due to long-term effects on the inflammatory lesions, higher incidence of gingival recession and others clinical parameters in smokers is correlated with cytotoxic and vasoactive substances present in tobacco, including nicotine, carbon monoxide and reactive oxidant substances and systemic effect is that smoking is responsible for 90% of cases of lung cancer, type deadliest cancer for men and women smokers, as well as being associated with various lung diseases. Furthermore, they promote oxidative stress and alterations in the immunoinflammatory responses, reducing functional activity of leucocytes, macrophages, lymphocytes and other immune cells, impaired wound healing and microbial recognition.

Nonsurgical therapy using scaling and root planning is the most usual periodontal therapy, well-recognized by the improvement in clinical and microbiological parameters. Fewer studies evaluated longitudinal clinical and microbiological status of smokers undergoing periodontal maintenance therapy and controversial results were found with absence of difference in disease progression in comparison with nonsmokers. P. gingivalis has been reduced after periodontal treatment. Previous report related reduction of 93 % to P.gingivalis for non-smokers and 88 % for smokers after periodontal treatment.

ELIGIBILITY:
Inclusion Criteria:

Clinical diagnosis of chronic periodontitis Consumption of 10 or more cigarettes/day.

Exclusion Criteria:

Diabetes mellitus Osteoporosis Pregnant and lactating females Immune suppressive medication Phenytoin Cyclosporine Calcium channel blockers Immunotherapy or diagnosed as HIV+

Ages: 27 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2016-08; Primary Completion 2016-10 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
Change from baseline Bleeding on Probe to 3 months | 3 months
  Bleeding On Probe will be expressed in percentage per individual to evaluate presence of bleeding on probe.
Change from Baseline Plaque Index to 3 months | 3 months
  Plaque Index will be expressed in percentage per individual to evaluate presence of plaque.
Change from Baseline Pocket Probing Depth to 3 months | 3 months
  Pocket Probing Depth will be evaluated in millimeter. The measure will be performed at six sites per tooth using a periodontal probe.
Change from Baseline Gingival Recession to 3months | 3 months
  Gingival Recession will be evaluated in millimeter. The measure will be performed at six sites per tooth, from cementoenamel junction to gingival margin, using a periodontal probe.
Change from Baseline Clinical Attachment level to 3 months | 3 months
  Clinical Attachment Level will be evaluated in millimeter. The measure will be performed at six sites per tooth, from cementoenamel junction to the end of periodontal pocket, using a periodontal probe.
Change from Baseline Biofilm to 3 months | 3 months
  Pooled biofilms from each site with Probe Depth >5mm will be collected and checked for the presence of fimbrial subunit genotype of Porphyromonas gingivalis I, II, III, IV and V by Polymerase Chain Reaction analysis. The results will be expressed by percentage of frequency of each type of fim A.
Change from baseline Age to 3 months | 3 months
  Age will be expressed in years.
Change from Baseline Cigarette consumption to 3 months | 3 months
  Time of cigarette consumption - will be expressed in years.

IPD SHARING:
Plan to Share IPD: Yes
The result will be communicated verbally for each participant.

REFERENCES:
- [Result] Lin X, Wu J, Xie H. Porphyromonas gingivalis minor fimbriae are required for cell-cell interactions. Infect Immun. 2006 Oct;74(10):6011-5. doi: 10.1128/IAI.00797-06. PMID 16988281
- [Result] Zhao L, Wu YF, Meng S, Yang H, OuYang YL, Zhou XD. Prevalence of fimA genotypes of Porphyromonas gingivalis and periodontal health status in Chinese adults. J Periodontal Res. 2007 Dec;42(6):511-7. doi: 10.1111/j.1600-0765.2007.00975.x. PMID 17956463
- [Result] Amano A, Kuboniwa M, Nakagawa I, Akiyama S, Morisaki I, Hamada S. Prevalence of specific genotypes of Porphyromonas gingivalis fimA and periodontal health status. J Dent Res. 2000 Sep;79(9):1664-8. doi: 10.1177/00220345000790090501. PMID 11023261
- [Result] Zeller I, Hutcherson JA, Lamont RJ, Demuth DR, Gumus P, Nizam N, Buduneli N, Scott DA. Altered antigenic profiling and infectivity of Porphyromonas gingivalis in smokers and non-smokers with periodontitis. J Periodontol. 2014 Jun;85(6):837-44. doi: 10.1902/jop.2013.130336. Epub 2013 Oct 23. PMID 24147843